CLINICAL TRIAL: NCT00558298
Title: Risperidone Depot (Microspheres) in the Treatment of Subjects With Schizophrenia or Schizoaffective Disorder - an Open Label Follow up Trial of RIS-INT-57 and RIS-INT-61.
Brief Title: A Long Term Study of Safety for Long Acting Injectable Risperidone in Patients With Schizophrenia or Schizoaffective Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CR002023
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; risperidone; intramuscular injection; long-acting injectable
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to document the long-term safety of 25, 50 or 75 mg long-acting injectable risperidone given via injection to the gluteal muscle every 2 weeks to patients with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Noncompliance in taking medication is very common among people with schizophrenia, and is a frequent cause of relapse of symptoms. A long-acting injectable formulation that ensures the slow but steady release of risperidone over a period of several weeks would eliminate the need to take medication on a daily basis, and improve compliance. This is an open-label, international, multicenter study in patients with schizophrenia or schizoaffective disorder who either completed study RIS-INT-57 or RIS-INT-61 or who dropped out of RIS-INT-61 after the completion of 3 injection cycles. Patients have to begin this study within 7 days of the final endpoint visit in the RIS-INT-57 or RIS-INT-61 studies. The endpoint visit of RIS-INT-57 and RIS-INT-61 serves as the first visit (Visit 1) of RIS-INT-63, and is considered the baseline of this extension study. Patients who have completed RIS-INT-57 will continue to receive the same dose of long-acting injectable risperidone (25, 50 or 75 mg) as they received during the last 3 months of that study. Patients who have completed or dropped out of RIS-INT-61 will continue to receive the same or equivalent dose of long-acting injectable risperidone as they had received during that study. The blind will not be broken for patients from the RIS-INT-61 study, therefore they will continue to receive double-blind oral medication for the first 3 weeks of this extension study. The total study duration is planned to be at least 1 year. The study hypothesis is that treatment with the long-acting injectable formulation of risperidone every 2 weeks for at least 1 year will be safe and well tolerated, as assessed by adverse event reporting, the extrapyramidal symptom rating scale, laboratory tests, vital signs measurements, physical examinations, body weight measurements, electrocardiograms, and injection site evaluations. Patients will receive injections of risperidone depot in microspheres (25, 50 or 75 mg) in their muscle at 2-weekly intervals for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (patients from RIS-INT-57 or RIS-INT-61) or schizoaffective disorder (patients from RIS-INT-57 only) according to the DSM-IV criteria
* patient completed RIS-INT-57 or RIS-INT-61 or dropped out after completion of 3 injection cycles in RIS-INT-61 (i.e., at or after Visit 4)
* Patient was otherwise healthy on the basis of a prestudy physical examination and medical history.

Exclusion Criteria:

* No DSM-IV diagnosis of substance abuse or dependence within 3 months prior to entry in RIS-INT-57 or RIS-INT-61 (excluding nicotine and caffeine dependence)
* No pregnant or breast-feeding women
* No female patient of childbearing potential without adequate contraception
* No history of severe drug allergy or hypersensitivity
* No patients known to be unresponsive to risperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2000-02; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To document the long-term safety of 25, 50 and 75 mg long-acting injectable risperidone from baseline until study endpoint.

SECONDARY OUTCOMES:
The mean values and change from baseline in Clinical Global Impression scale (CGI) at each time point until study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- See also: A long term safety study for long acting injectable risperidone in schizophrenia or schizoaffective disorder patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=344&filename=CR002023_CSR.pdf